CLINICAL TRIAL: NCT06223412
Title: Video-Based Climate Change Program on Revitalizing Eco-Cognizance, Emotional Response, and Self-efficacy Among Nursing Students in Rural Communities: A Randomized Controlled Study
Brief Title: Video-based Climate Change Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19102023
Record Dates: First submitted 2023-12-23; First posted 2024-01-25 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Anxiety State; Efficacy, Self
Keywords: Awareness, Emotion, Self-efficacy, Climate change.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): The participants in this group received a series of short videos, ranging between 30- 45 minutes/ each video revolved around five core themes including The road start to green planet, The ripple effect climate change on Health, Climate Change Literacy, Strengthen resilience to overcome climate related- psychological impacts, and Sustaining phase: closing session..
  Interventions: Behavioral: video-based climate change program
- control group (Placebo Comparator): The participants in this group received routine care such as received flyers related to climate change across the globe.
  Interventions: Behavioral: video-based climate change program

INTERVENTIONS:
Behavioral: video-based climate change program — The participants in this group received a series of short videos, ranging between 30- 45 minutes/ each video revolved around five core themes including The road start to green planet, The ripple effect climate change on Health, Climate Change Literacy, Strengthen resilience to overcome climate related- psychological impacts, and Sustaining phase: closing session.

SUMMARY:
Climate change represents a global crisis with far-reaching implications for health, including mental health. Among vulnerable populations, such as nursing students, climate change anxiety is emerging as a noteworthy concern. Recognizing the need to address this issue, our research aims to investigate the impact of a virtual-based program on climate change awareness, anxiety levels, and self-efficacy among nursing students. As future healthcare professionals, nursing students play a pivotal role in promoting sustainable health practices and addressing the health impacts of climate change. This study seeks to contribute valuable insights into the effectiveness of virtual interventions in raising awareness and enhancing the coping mechanisms of nursing students in the face of climate change challenges.

DETAILED DESCRIPTION:
Aim:

to investigate the effect of a video-based climate change program on revitalizing eco-cognizance, emotional response, and self-efficacy among nursing students in rural communities when compared to a group who received flyers related to climate change across the globe.

Research Hypothesis

* Hypothesis 1: The video-based climate change program will significantly improve climate change perceptions among college students in rural communities.
* Hypothesis 2: The video-based climate change program will significantly improve environmental self-efficacy among college students in rural communities.
* Hypothesis 3: The video-based climate change program will significantly reduce climate change anxiety among college students in rural communities.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, students had to be from 2nd academic year to 4th year, not enter any educational program about climate change, owning a smartphone, and willingness to participate in program.

Exclusion Criteria:

* students who have psychological problems

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Climate change perceptions | 1 month
  Climate change perceptions was developed to examine participants' views on the reality, causes, and outcomes of climate change. Respondents rated each 14 item on a 7-point scale, ranging from completely disagree to completely agree.

SECONDARY OUTCOMES:
Environmental self-efficacy scale (ESE) | 1 month
  Environmental self-efficacy scale (ESE) developed by Bryton & Alexander (2019). It is used to measure environmental self-efficacy. It consists of 20 items rated on a 11-point Likert scale, with 0 denotes cannot do at all, and 10 denotes highly certain can do, with higher scores indicating higher environmental self-efficacy.
Climate Change Anxiety Scale | 1 month
  The Climate Change Anxiety Scale, developed by Clayton and Karazsia in 2020, is a specialized instrument designed to measure the psychological distress associated with climate change. Comprising 13 items, respondents rate each item on a scale ranging from 1 (never) to 5 (almost always).

CONTACTS AND LOCATIONS:
Overall Officials: rasha eweida, Study Chair — Damanhour University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toan do TT, Kien VD, Bao Giang K, Van Minh H, Wright P. Perceptions of climate change and its impact on human health: an integrated quantitative and qualitative approach. Glob Health Action. 2014 Dec 8;7:23025. doi: 10.3402/gha.v7.23025. eCollection 2014. PMID 25511880
- [Background] van Baal K, Stiel S, Schulte P. Public Perceptions of Climate Change and Health-A Cross-Sectional Survey Study. Int J Environ Res Public Health. 2023 Jan 13;20(2):1464. doi: 10.3390/ijerph20021464. PMID 36674220
- [Derived] Eweida RS, O'Connell MA, Zoromba M, Mahmoud MF, Altheeb MK, Selim A, Atta MHR. Video-Based Climate Change Program Boosts Eco-Cognizance, Emotional Response and Self-Efficacy in Rural Nursing Students: Randomised Controlled Trial. J Adv Nurs. 2025 Dec;81(12):8371-8383. doi: 10.1111/jan.16790. Epub 2025 Mar 9. PMID 40059412